CLINICAL TRIAL: NCT02356445
Title: Outcome of Use of Cytotoxic Drugs for Inflammatory Lung Diseases
Brief Title: Use of Immunosuppressive Therapy for Sarcoidosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Robert P Baughman, Professor of Medicine, University of Cincinnati
Other Study IDs: UCincinnati
Record Dates: First submitted 2014-11-03; First posted 2015-02-05 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Cytotoxins; Methotrexate; Azathioprine; Infliximab; Adrenocorticotropic Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum in some cases
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cytotoxic drug: Patients treated for sarcoidosis
  Interventions: Other: Cytotoxic drug

INTERVENTIONS:
Other: Cytotoxic drug — Observe patients versus treatment type
  Other Names: Methotrexate, azathioprine, infliximab, Acthar

SUMMARY:
Retrospective review of the outcome of use of immunosuppressive drugs in treatment of sarcoidosis

DETAILED DESCRIPTION:
Patients receiving one or more cytotoxic or other immunosuppressive drug will be observed

ELIGIBILITY:
Inclusion Criteria:

Any patient treated for sarcoidosis

Exclusion Criteria:

* None

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with sarcoidosis treated
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcome | 2 years
  Number of participants with improvement over two years

SECONDARY OUTCOMES:
Toxicity | 2 years
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Baughman, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Baughman RP, Kotzin J, Lower EE. The Value of a Patient Global Assessment in Management of Sarcoidosis. Lung. 2021 Aug;199(4):357-362. doi: 10.1007/s00408-021-00455-5. Epub 2021 Jul 13. PMID 34255140
- [Derived] Zhou Y, Lower EE, Li HP, Costea A, Attari M, Baughman RP. Cardiac Sarcoidosis: The Impact of Age and Implanted Devices on Survival. Chest. 2017 Jan;151(1):139-148. doi: 10.1016/j.chest.2016.08.1457. Epub 2016 Sep 8. PMID 27614001